CLINICAL TRIAL: NCT03020641
Title: Characterization of Changes in Peritoneal Cells Gene Expression After Standard Versus Low Pressure Laparoscopic Cholecystectomy and Its Clinical Correlation
Brief Title: Peritoneal Damage in Laparoscopic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacion para la Investigacion Biomedica del Hospital Universitario Ramon y Cajal (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: A-CGyD-2017
Record Dates: First submitted 2017-01-09; First posted 2017-01-13 (Estimated); Results first posted 2021-09-22 (Actual); Last update posted 2021-09-22 (Actual); Status verified 2021-09

CONDITIONS: Peritoneal Damage
Keywords: low pressure pneumoperitoneum; standard pressure pneumoperitoneum; laparoscopy cholecystectomy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low pneumoperitoneum pressure. (Experimental): Pneumoperitoneum pressure at 8 mmHg or lower.
  Interventions: Procedure: Low pressure pneumoperitoneum
- standard pneumoperitoneum pressure (Active Comparator): Pneumoperitoneum pressure at 12 mmHG or higher
  Interventions: Procedure: standard pneumoperitoneum pressure

INTERVENTIONS:
Procedure: Low pressure pneumoperitoneum — Low pressure pneumoperitoneum
  Arms: Low pneumoperitoneum pressure.
Procedure: standard pneumoperitoneum pressure — standard pneumoperitoneum pressure
  Arms: standard pneumoperitoneum pressure

SUMMARY:
The investigators hypothesized that applying a low intraperitoneal pressure pneumoperitoneum (≤ 8mmHg) during laparoscopic cholecystectomy, the adverse impact on the surgical peritoneal environment (measured as gene expression of extracellular matrix, adhesion and inflammatory cytokine as well as oxidative stress response and apoptotic index), can be minimized and probably clinical outcomes might be better.

DETAILED DESCRIPTION:
Cholelithiasis is one of the most frequent abdominal diseases requiring surgical treatment. Laparoscopic cholecystectomy is currently the procedure of choice to remove the gallbladder. There is growing evidence that increased intra-abdominal pressure pneumoperitoneum, even for short periods of time, is associated with both transient and sometimes persistent adverse effects that might negatively affect the surgical peritoneal environment .There are some studies that have demonstrated that using low intraperitoneal pressure pneumoperitoneum, undesired effects like adverse impact on peritoneal tissue and negative clinical outcomes could be reduced.Therefore intraperitoneal pressure target during laparoscopy should be the lowest to allow surgery be securely performed. Many strategies have been tested in order to improve the volume of gas can be insufflated inside the abdominal cavity while maintaining low pneumoperitoneum pressure during laparoscopy.So far the most studied strategy has been deep neuromuscular blockade.However the effect of the depth of neuromuscular blockade in the intraabdominal volume is still controversial as sometimes in humans its benefits are marginal.There is scarce information in the medical literature regarding the adverse impact on peritoneal tissue of high pneumoperitoneum pressure during laparoscopy in humans. In addition available data are provided by non-prospective, non-randomized and small sample studies, so randomized controlled trials are required to ascertain this issues.To our knowledge our study is the first prospective and randomized controlled trial in humans aiming to study the adverse impact of high pressure pneumoperitoneum on peritoneal tissue as well as to associate it with clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years, signed informed consent, undergoing laparoscopic cholecystectomy for symptomatic cholelithiasis or gallbladder polyps.

Exclusion Criteria:

* Emergency surgery.
* Previous surgery at supramesocolic compartment.
* Previous peritoneal inflammatory process.
* Pregnancy or breastfeeding.
* Patient refusal to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2017-01-27 (Actual); Primary Completion 2019-04-28 (Actual); Study Completion 2019-04-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Ramon y Cajal Hospital, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Data were collected from January 2017 to May 2019
Groups:
- Control: Standard pneumoperitoneum pressure (12 mmHg or lower) during laparoscopic cholecystectomy to evaluate the peritoneal tissue damage
- Intervention: Low pneumoperitoneum pressure (8 mmHg or lower) during laparoscopic cholecystectomy to evaluate the peritoneal tissue damage
Period: Overall Study
Arm/Group | Control | Intervention
Started | 50 | 50
Completed | 48 | 47
Not Completed | 2 | 3
Not completed — Lost to Follow-up | 0 | 1
Not completed — Converted to open surgery | 2 | 1
Not completed — for surgery not performed | 0 | 1

BASELINE CHARACTERISTICS:
Population: 5 patients were excluded see Participant flow for more details
Groups:
- Experimental: Low pneumoperitoneum pressure (8 mmHg or lower) during laparoscopic cholecystectomy to evaluate the peritoneal tissue damage
- Total: Total of all reporting groups
Arm/Group | Experimental | Control | Total
Number analyzed (Participants) | 47 | 48 | 95
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.47 (16.88) | 51.71 (15.72) | 53.04 (16.26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 37 | 69
  Male | 15 | 11 | 26
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
BMI [Mean (Standard Deviation); unit: kg/m^2] — Body mass index
  kg/m^2 | 26.63 (4.07) | 27.51 (4.6) | 27.07 (4.3)
ASA [Count of Participants; unit: Participants] — American Society Anaesthesiologists classification. ASA I A normal healthy patient ASA II A patient with mild systemic disease ASA III A patient with severe systemic disease ASA IV A patient with severe systemic disease that is a constant threat to life ASA V A moribund patient who is not expected to survive without the operation ASA VI A declared brain-dead patient whose organs are being removed for donor purposes
  Participants
    I | 16 | 12 | 28
    II | 23 | 32 | 55
    III | 7 | 4 | 11
    IV | 0 | 0 | 0
    Unknow | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Inflammatory Peritoneal Markers
Description: logaritmic levels of mRNA of the different markers at time 1 hour after creation of the pneumoperitoneum
Time Frame: he values will be obtained from the study of peritoneal tissue samples one hour after the creation of the pneumoperitoneum (T1).
Population: 23 excluded samples
Measure: Mean (Standard Deviation); unit: log (pg/ml)
Arm/Group | Control | Experimental
Number analyzed (Participants) | 40 | 37
log (pg/ml)
  Interleukin 1 | 0.80 (1.00) | 1.14 (1.06)
  Interlerukin 6 | 4.26 (1.34) | 3.24 (1.21)
  Interleukin 10 | 0.76 (1.01) | 1.10 (0.84)
  vascular endotelial growth factor A | 0.09 (0.99) | -0.05 (0.50)
  Tumor necrosis factor α | -0.71 (0.99) | -0.74 (0.71)
  CXC lingand 2 | 2.18 (0.99) | 2.22 (0.72)
Statistical Analysis 1: Comparison: Control vs Experimental; Interleukin 1 (IL1); Test type: Other — t-test; p = 0.058, t-test, 2 sided — the threshold for statistical significance was p<=0.05; Mean Difference (Net) = - 0.34, 95% CI 2-sided [- 0.8077 to 0.1276], Standard Error of Mean 0.2347
Statistical Analysis 2: Comparison: Control vs Experimental; Test type: Other — Interleukin 6 (IL6); p = 0.001, t-test, 2 sided; Mean Difference (Final Values) = -1.02, 95% CI 2-sided [-1.60 to -0.44], Standard Error of Mean 0.29
Statistical Analysis 3: Comparison: Control vs Experimental; Interleukin 10; Test type: Other; p = 0.052, t-test, 2 sided; Mean Difference (Net) = 0.34, 95% CI 2-sided [-0.76 to 0.81], Standard Error of Mean 0.211
Statistical Analysis 4: Comparison: Control vs Experimental; Vascular Endotelial Grow Factor A; Test type: Other; p = 0.815, t-test, 2 sided; Mean Difference (Final Values) = -0.14, 95% CI 2-sided [-0.50 to 0.22], Standard Error of Mean 0.181
Statistical Analysis 5: Comparison: Control vs Experimental; TNF alfa; Test type: Other; p = 0.742, t-test, 2 sided; Mean Difference (Final Values) = -0.03, 95% CI 2-sided [-0.42 to 0.36], Standard Error of Mean 0.19
Statistical Analysis 6: Comparison: Control vs Experimental; Chemokine CXC ligand 2; Test type: Other; p = 0.603, t-test, 2 sided; Mean Difference (Final Values) = 0.04, 95% CI 2-sided [-0.36 to 0.44], Standard Error of Mean 0.2

2. Primary Outcome: Remodeling Peritoneal Markers :( Gene Expression (mRNA) Levels of)
Description: f. CTGF "connective tissue growth factor". g. MMP-9 "matrix metalloproteinase-9". h. PAI-I "plasminogen activator inhibitor-I". i. E-selectin. Samples will be processed to obtain total RNA with TRI Reagent™ (Sigma) and will be quantified with NanoDrop spectrophotometer.
Time Frame: The values will be obtained from the study of peritoneal tissue samples one hour after the creation of the pneumoperitoneum (T1).
Population: 13 samples excluded
Measure: Mean (Standard Error); unit: log (pg/ml)
Arm/Group | Intervention | Control
Number analyzed (Participants) | 37 | 40
log (pg/ml)
  Connective tissue growth factor | 0.89 (0.61) | 0.61 (0.84)
  Matrix metalloproteinasa-9 | 0.56 (1.15) | 0.47 (1.31)
  Plasminogenin activator inhibitor | 0.74 (0.89) | 0.24 (1.15)
  E- selectin | 0.66 (139) | 0.57 (1.77)
Statistical Analysis 1: Comparison: Intervention vs Control; Matrix metalloproteinase-9; Test type: Other; p = 0.600, t-test, 2 sided; Mean Difference (Final Values) = 0.09, 95% CI 2-sided [-0.47 to 0.65], Standard Error of Mean 0.28
Statistical Analysis 2: Comparison: Intervention vs Control; Plasminogen activator inhibitor-1; Test type: Other; p = 0.028, t-test, 2 sided; Mean Difference (Final Values) = 0.50, 95% CI 2-sided [0.030 to 0.97], Standard Error of Mean .24
Statistical Analysis 3: Comparison: Intervention vs Control; E-selectin; Test type: Other; p = 0.807, t-test, 2 sided; Mean Difference (Final Values) = 0.09, 95% CI 2-sided [-0.64 to 0.82], Standard Error of Mean 0.36

3. Primary Outcome: Oxidative Stress Response Marker:MDA (Malondialdehyde)
Description: MDA (malondialdehyde) determination will be done with ELISA
Time Frame: The values of the main variables will be obtained from the study of peritoneal tissue samples one hour after the creation of the pneumoperitoneum (T1)
Population: It was impossible to measure MDA due to laboratory problems.
Arm/Group | Experimental | Control
Number analyzed (Participants) | 0 | 0

4. Primary Outcome: Apoptotic Index
Description: This measure is reported as the mean of the difference of the percentage of apoptotic cells at baseline minus the final
Time Frame: The values of the main variables will be obtained from the study of peritoneal tissue samples, one hour after the creation of the pneumoperitoneum compared to basal peritoneal tissue samples.
Population: 13 samples excluded
Measure: Mean (Standard Deviation); unit: difference of the percentage
Arm/Group | Control | Experimental
Number analyzed (Participants) | 40 | 37
difference of the percentage | -1.92 (24.3) | -0.56 (12.3)
Statistical Analysis 1: Comparison: Control vs Experimental; Test type: Other; p = 0.862, t-test, 2 sided; Mean Difference (Final Values) = -1.37, 95% CI 2-sided [-7.49 to 10.21], Standard Error of Mean 4.44

ADVERSE EVENTS:
Time Frame: no adverse event data. All-Cause Mortality, Serious, and Other [Not Including Serious] Adverse Events were not monitored/assessed."
Description: All-Cause Mortality, Serious, and Other [Not Including Serious] Adverse Events were not monitored/assessed."
Arm/Group | Control | Experimental
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
no limitations

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-27): https://cdn.clinicaltrials.gov/large-docs/41/NCT03020641/Prot_SAP_000.pdf